CLINICAL TRIAL: NCT05185128
Title: Neural Basis of Social Cognition Deficits in Youth With Autism and Schizophrenia
Brief Title: Neural Basis of Social Cognition Deficits
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5200189
Record Dates: First submitted 2021-12-23; First posted 2022-01-11 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Autism Spectrum Disorder; Psychosis; Social Communication
MeSH Terms: conditions — Autism Spectrum Disorder; Psychotic Disorders; Communication

STUDY DESIGN:
Intervention Model Description: The PEERS treatment program consists of 90-minute sessions, delivered once a week over the course of 16- weeks. Parents and children/adolescents attend separate concurrent sessions that instruct them on key elements about making and keeping friends. Participants in both the ASD and SSD groups will engage in approximately three hours of diagnostic, behavioral, and social cognition testing and one hour of MRI scanning both pre- and post-treatment. Additionally, TD participants will undergo two MRI scanning and behavioral assessment sessions approximately 16-weeks apart without enrolling in the PEERS program, to serve as controls.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): Typically developing control participants will undergo cognitive assessments and MRI imaging 16 weeks apart with no intervention in between.
- Patient arm (Experimental): Both ASD and SSD participants will undergo cognitive assessments and MRI imaging pre- and post- the 16-week PEERS social skills intervention.
  Interventions: Behavioral: PEERS social skills intervention

INTERVENTIONS:
Behavioral: PEERS social skills intervention — The PEERS treatment program consists of 90-minute sessions, delivered once a week over the course of 16- weeks. Parents and children/adolescents attend separate concurrent sessions that instruct them on key elements about making and keeping friends. Among others, this parent-assisted, social skills intervention provides explicit instruction to target verbal and nonverbal communication skills, appropriate use of humor and resolving peer conflict, as well as expanding and developing friendship networks38. The candidate, Dr. Nair, has been trained on the PEERS social skills intervention extensively for the past five years, and is a certified provider for the adolescent program. The PEERS program will be provided by Dr. Nair's research team (consisting of Dr. Nair, lab co-ordinators, and clinical psychology doctoral students) through the LLU Department of Psychology.
  Arms: Patient arm

SUMMARY:
Difficulties in reciprocal social interaction are hallmark features of several neuropsychiatric disorders, most notably autism spectrum disorder (ASD) and schizophrenia spectrum disorder (SSD). While recent studies have demonstrated substantial overlap in genetic etiology between ASD and SSD, little is known about common versus unique neural mechanisms that may underlie these downstream social deficits that cross diagnostic boundaries. Thus, a comprehensive imaging study examining social deficits in youth with ASD and adolescent- onset SSD at the neurochemical, connectivity, as well as functional activation level will be crucial in furthering our understanding of these underlying neural mechanisms. Specifically, the current project aims to examine how targeted social skills interventions may impact the organization of large-scale functional brain networks implicated in social cognition in these disorders, leading to improved outcomes. Thirty adolescents with ASD and 30 adolescents with SSD will undergo the Program for the Education and Enrichment of Relational Skills (PEERS), which is a 16-week parent-assisted social skills intervention that aims to improve friendship quality and social skills in teens with social difficulties. All participants will receive pre- and post-treatment MRI scans including functional MRI and magnetic resonance spectroscopy to quantify neural changes resulting from the intervention. All participants will also receive behavioral and social cognition assessments pre- and post-intervention to quantify real- world gains in social behaviors resulting from the intervention. Additionally, 30 typically developing adolescents will be recruited to serve as control participants and undergo two MRI and behavioral assessment sessions 16-weeks apart with no intervention in between. Specific aims include (1) examining inter-group disruptions in connectivity patterns, activation levels, and neurometabolite concentrations in key social brain regions pre-treatment in ASD and SSD groups, (2) examining inter-group changes in connectivity patterns, activation levels, and neurometabolite concentrations in key social brain regions in response to treatment in ASD and SSD groups, and, (3) dimensionally identifying intra-group differences in brain responses and how they relate to real-world treatment outcomes.

DETAILED DESCRIPTION:
Difficulties in reciprocal social interaction are hallmark features of several neuropsychiatric disorders, most notably autism spectrum disorder (ASD) and schizophrenia spectrum disorder (SSD). Recent behavioral studies of adults with SSD and ASD have highlighted not only the similarities but also some divergent patterns of social impairments in the two disorders - with ASD characterized by lower social motivation, poorer social reciprocity, and undermentalizing, and SSD characterized by greater reciprocity but poor expressiveness. Given the public health significance of social disability and social isolation, it is crucial to explore the neurobiological mechanisms underlying these social skill deficits across both groups, as well as to understand how these relate to real-world behaviors. Although antipsychotics have been shown to be effective in reducing positive symptoms in SSD, they are not effective in addressing the devastating social disability associated with the disorder, which contributes to chronic functional impairment. It is thus imperative to identify behavioral interventions for children and adolescents that have already shown promise in other clinical groups such as ASD. By enhancing our understanding of the neurobiological underpinnings of social impairments in adolescent-onset SSD and how they compare to those observed in ASD, we will be able to refine treatment targets and better predict outcomes for each group. To this effect, the proposed study will examine biomarkers that are likely related to positive outcomes from targeted social skills intervention in adolescents with SSD and ASD. Building upon an established evidence-based treatment - the Program for the Education and Enrichment of Relational Skills (PEERS), we will collect resting state functional imaging (rs-fcMRI), task-paradigm functional BOLD activation (fMRI), and magnetic resonance spectroscopy (MRS) before and after 30 SSD and 30 ASD adolescents, 12-18 years of age, undergo the 16-week evidence-based PEERS behavioral intervention. These data will then be compared to a matched sample of 30 typically developing (TD) adolescents who are not enrolled in the PEERS program but will undergo two MRI scans 16-weeks apart. The overarching goal of the study will be to create a novel multimodal neuroimaging design to examine the neural underpinning of social difficulties in SSD and ASD, explore neuroplasticity in both groups in response to a brief targeted social-skills intervention, and predict treatment response and its contribution to long-term maintenance of skills after treatment completion.

The following are the study's specific aims:

Aim 1: Assess treatment related changes in 'social brain' regions following evidence-based social skills training in ASD and SSD group, compared to neural patterns observed in TD adolescents.

Hypothesis 1a: rs-fcMRI indices within social brain networks will look more improved (similar to TD adolescents) post-treatment compared to pre-treatment for the both ASD and SSD groups (e.g., greater connectivity in social brain networks in ASD group, lower connectivity of extraneous regions in SSD group).

Hypothesis 1b: fMRI brain activation in social brain regions in response to the social task-paradigm will look more improved (similar to TD adolescents) post-treatment compared to pre-treatment for both ASD and SSD group (e.g., greater activation in social brain networks in ASD group, lower activation of extraneous regions in SSD group). Hypothesis 1c: There will be significant improvement (similar to TD adolescents) in MRS indices of GABA (inhibitory) and glutamate (excitatory) neurometabolite concentrations within social brain networks in ASD and SSD post- treatment compared to pre-treatment (e.g., lower glutamate/higher GABA in social brain regions in ASD group, higher glutamate/higher GABA in social brain regions in SSD group).

Aim 2: To test whether pre- and post-treatment neural changes are meaningfully related to behavioral measures of treatment outcome.

Hypothesis 2: Neural responses post-intervention will correlate with gains in social motivation and reciprocity behavioral outcomes measures in the ASD group, and gains in social expressivity outcome measures in the SSD group.

Exploratory Aim 3: Given that both ASD and SSD are characterized as spectrum disorders of varying severity, heterogeneous etiologies, and comorbidities, we aim to explore how individual differences in patterns of brain connectivity and activation might predict treatment response and treatment maintenance dimensionally in addition to the category-based diagnostic systems proposed above. Given the exploratory nature of the proposed aim, specific hypotheses are not projected regarding the precise changes in neural activity on an individual basis. However, accomplishing this goal will us understand underlying neural mechanisms of treatment-related change across groups, and serve to better target interventions to address the heterogeneity of social cognition deficits observed in both ASD and SSD.

ELIGIBILITY:
Inclusion Criteria:

Participants in this study will be 30 ASD adolescents and 30 demographically matched adolescents with SSD who undergo the PEERS social skills training program. Participants will be between the ages of 12-18 years, and mostly male reflecting the higher prevalence in the population of ASD, and to a lesser extent, SSD. The ASD adolescents will be recruited through the Loma Linda University Behavioral Health Institute (LLU BHI), LLU Behavior Medicine Center (BMC), and LLU Department of Psychology Child and Family Center (CFC). The SSD adolescents will be recruited from the BMC inpatient, partial hospitalization, intensive outpatient, and standard outpatient programs for youth with psychosis. Thirty demographically comparable typically developing (TD) controls will be recruited through community samples, and in compliance with the LLU Institutional Review Board (IRB) standards. Before enrolling in the proposed MRI studies, prospective ASD participants will undergo testing with experienced assessors. Clinical diagnosis will be confirmed using both the Autism Diagnostic Interview- Revised, and the Autism Diagnostic Observation Schedule, 2nd edition. SSD participants will be screened using the Structured Clinical Interview for DSM-IV (SCID) Axis I diagnoses, with additional modules for assessment of childhood disorders. SSD participants must meet criteria for schizophrenia, schizophreniform, schizoaffective disorder, or unspecified schizophrenia spectrum and other psychotic disorder. All study participants will have verbal IQ as well as Full Scale IQ of 70 or higher on the Wechsler Abbreviated Scale of Intelligence (WASI-II) to ensure they will have the language and cognitive ability to participate in an MRI scan.

Exclusion Criteria:

Exclusion criteria will include history of significant medical/neurologic conditions that would affect neuroimaging interpretation (e.g., epilepsy, tumor), and any psychiatric history for TD controls. Participants with any MRI contraindications (e.g., history of metal fragment injury or metal implants, current orthodontic braces or nonremovable retainers) will also be excluded in compliance with scanner safety standards.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The Awareness of Social Inference Test (TASIT) | Change between baseline and final visit at week 16
  This is a Theory of Mind (ToM) measure containing 16 videotaped scenes. After each scene, subjects respond to questions about the characters' intentions, beliefs about the situation, and emotional state.
The Social Attribution Task - Multiple Choice (SAT-MC, SAT-MC-II) | Change between baseline and final visit at week 16
  his test uses a 64- second video of geometric shapes set in motion to portray themes of social relatedness and intentions. Considered a test of "Theory of Mind," the SAT-MC and its alternative form SAT-MC-II assesses implicit social attribution formation while reducing verbal and basic cognitive demands.
The computerized Penn Emotion Identification Task (PennCNB) | Change between baseline and final visit at week 16
  The PennCNB Emotion Identification Test (EMI) measures the ability to correctly identify facial expressions of emotion. Participants are shown 40 faces one at a time on the computer, and must identify the emotion expressed by the actors face from multiple choice options provided.

SECONDARY OUTCOMES:
Functional MRI | Change between baseline and final visit at week 16
  rs-fcMRI indices within social brain networks will look more improved (similar to TD adolescents) post-treatment compared to pre-treatment for the both ASD and SSD groups (e.g., greater connectivity in social brain networks in ASD group, lower connectivity of extraneous regions in SSD group). Rate of connectivity ranges from -3 low to +3 high connectivity.

CONTACTS AND LOCATIONS:
Overall Officials: Aarti Nair, PhD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda U, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No